CLINICAL TRIAL: NCT01644253
Title: Phase 1b, Open Label Study to Evaluate Safety and Efficacy of TRU-016 in Combination With Rituximab, Obinutuzumab, Rituximab and Idelalisib, or Ibrutinib in Chronic Lymphocytic Leukemia and With Bendamustine in Peripheral T-cell Lymphoma
Brief Title: Phase 1b Safety and Efficacy Study of TRU-016
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Aptevo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16009
Record Dates: First submitted 2012-07-12; First posted 2012-07-19 (Estimated); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Chronic Lymphocytic Leukemia; Peripheral T-cell Lymphoma
Keywords: chronic lymphocytic leukemia; CLL; previously untreated chronic lymphocytic leukemia; peripheral T-cell lymphoma; PTCL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, T-Cell, Peripheral | interventions — TRU 016; Rituximab; obinutuzumab; idelalisib; ibrutinib; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort 1 - Previously Untreated CLL (Experimental): 20 mg/kg TRU-016 + Rituximab
  Interventions: Biological: 20 mg/kg TRU-016 + Rituximab
- Cohort 2 - Relapsed CLL (Experimental): 20 mg/kg TRU-016 + Rituximab
  Interventions: Biological: 20 mg/kg TRU-016 + Rituximab
- Cohort 3 - Previously Untreated CLL (Experimental): 10 mg/kg TRU-016 + Rituximab
  Interventions: Biological: 10 mg/kg TRU-016 + Rituximab
- Cohort 4 - Previously Untreated CLL (Experimental): 20 mg/kg TRU-016 20 + Obinutuzumab
  Interventions: Biological: TRU-016 20 mg/kg + Obinutuzumab
- Cohort 5 - Relapse CLL (Experimental): 20 mg/kg TRU-016 + idelalisib + rituximab
  Interventions: Biological: TRU-016 6-20 mg/kg + idelalisib + rituximab
- Cohort 6 - With CLL on ibrutinib with no complete response (Experimental): 20 mg/kg TRU-016 + ibrutinib
  Interventions: Biological: TRU-016 10-20 mg/kg + ibrutinib
- Cohort 7 - With CLL on ibrutinib with stable disease (Experimental): 20 mg/kg TRU-016 + ibrutinib
  Interventions: Biological: TRU-016 10-20 mg/kg + ibrutinib
- Cohort 8 - With relapsed or refractory PTCL (Experimental): 20 mg/kg TRU-016 + 90 mg/m2 bendamustine
  Interventions: Biological: TRU-016 10-20 mg/kg + bendamustine

INTERVENTIONS:
Biological: 20 mg/kg TRU-016 + Rituximab — TRU-016: 10 mg/kg for first dose, all subsequent doses 20 mg/kg, IV once weekly for 8 weeks followed by 4 monthly doses
  Rituximab: 375 mg/m2 for first dose, all subsequent doses 500 mg/m2, IV once weekly for 8 weeks followed by 4 monthly doses
  Other Names: Rituxan
  Arms: Cohort 1 - Previously Untreated CLL; Cohort 2 - Relapsed CLL
Biological: 10 mg/kg TRU-016 + Rituximab — TRU-016: 6 mg/kg for first dose, all subsequent doses 10 mg/kg, IV on Day 1, 8 and 15, followed by 5 monthly doses
  Rituximab: 375 mg/m2 for first dose, all subsequent doses 500 mg/m2, IV following TRU-016 schedule
  Other Names: Rituxan
  Arms: Cohort 3 - Previously Untreated CLL
Biological: TRU-016 20 mg/kg + Obinutuzumab — TRU-016: 6 mg/kg on Day 1, 20 mg/kg on Day 8 and 15, then 20 mg/kg once a month for 5 months
  Obinutuzumab: 100 mg on Day 1, 900 mg on Day 2, 1,000 mg on Day 8 and 15, then 1,000 mg once a month for 5 months
  Other Names: Gazyva
  Arms: Cohort 4 - Previously Untreated CLL
Biological: TRU-016 6-20 mg/kg + idelalisib + rituximab — TRU-016: 6 mg/kg on Days 15-36 weekly, 10 mg/kg on Days 43 and 50, then 20 mg/kg once a month for 5 months.
  Other Names: Zydelig, Rituxan
  Arms: Cohort 5 - Relapse CLL
Biological: TRU-016 10-20 mg/kg + ibrutinib — TRU-016: Dosed weekly for 8 weeks followed by 4 monthly intravenous (IV) infusions. The first dose will be 10 mg/kg and all subsequent doses will be 20 mg/kg.
  Other Names: Imbruvica
  Arms: Cohort 6 - With CLL on ibrutinib with no complete response; Cohort 7 - With CLL on ibrutinib with stable disease
Biological: TRU-016 10-20 mg/kg + bendamustine — TRU-016 dosed 10 mg/kg for the first dose and then 20 mg/kg weekly for 2 cycles, followed by dosing every other week for an additional 4 cycles (cycle = 28 days). Bendamustine (90 mg/m2 on days 2 and 3 of cycle 1 and then days 1 and 2 of cycles 2 to 6) will be infused after completion of TRU-016. If a patient is benefiting with stable disease or better, then TRU-016 may continue to be dosed every 3 weeks after the first 6 cycles; bendamustine will not be dosed beyond 6 cycles.
  Arms: Cohort 8 - With relapsed or refractory PTCL

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TRU-016 in combination with rituximab, in combination with obinutuzumab, in combination with rituximab and idelalisib, or in combination with ibrutinib in patients with CLL; and in combination with bendamustine in patients with PTCL.

DETAILED DESCRIPTION:
The study will consist of 8 dose cohorts:

1. Previously untreated patients 20 mg/kg TRU-016 + rituximab.
2. Relapsed patients, 20 mg/kg TRU-016 + rituximab.
3. Previously untreated patients 10 mg/kg TRU-016 + rituximab.
4. Previously untreated patients TRU-016 + obinutuzumab.
5. Relapsed patients, 20 mg/kg TRU-016 + rituximab + idelalisib.
6. Patients with CLL on ibrutinib or another BTK inhibitor for a total of more than 1 year who have not had a complete response (CR) will continue receiving ibrutinib or another BTK inhibitor.
7. Patients with CLL on ibrutinib or another BTK inhibitor with stable disease and in whom the cysteine 481 mutant clone is present at a level >1%, will continue receiving ibrutinib or the alternative BTK inhibitor.
8. Patients with relapsed or refractory PTCL will receive TRU-016 dosed 10 mg/kg for the first dose and then 20 mg/kg weekly for 2 cycles, followed by dosing every other week for an additional 4 cycles (cycle = 28 days) + bendamustine for 2 days every cycle for 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL by 2008 IWCLL criteria and with Rai stage intermediate or high risk CLL. Cohort 8 patients must have a diagnosis of PTCL.
* No prior therapy for CLL for Cohorts 1, 3 and 4. For Cohort 2, 1-3 prior treatments. For Cohort 5, patients must have failed to respond or relapsed after 1 or more treatment regimens. For Cohort 6, patients who have been receiving ibrutinib for at least 12 months, have not had a CR, and in whom no cysteine 481 mutation is detected. For Cohort 7, patients who are receiving ibrutinib with stable disease and now have the cysteine 481 mutant clone present at levels of >1%. For Cohort 8, have refractory or relapsed PTCL after one or more prior therapies.
* At least one of the following criteria for active disease requiring treatment: progressive splenomegaly and/or lymphadenopathy; anemia or thrombocytopenia due to bone marrow involvement; or progressive lymphocytosis with an increase of >50% over a 2-month period or an unanticipated doubling time of less than 6 months
* For Cohorts 1, 3 and 4, contraindication to chemotherapy as first-line therapy due to patient age, comorbidity or patient preference
* Age >/= to 18 years
* ECOG performance status of </= 2
* Life expectancy > 6 months in opinion of Investigator
* Serum creatinine, total bilirubin, ALT/SGPT </= 2.0 x upper limit of normal
* ANC >/= 800/mm3, Cohort 8 (PTCL): ANC >/= 1000/mm3
* Platelets >/= 30,000/mm3

Exclusion Criteria:

* For Cohorts 1, 3 and 4 only: Has received treatment with rituximab, alemtuzumab, ofatumumab or any other chemotherapeutic agent for CLL. Cohort 8: Received prior treatment with bendamustine and did not respond during treatment or relapsed less than sex months after completing treatment.
* Has received an investigational therapy within 30 days of first dose of study drug
* Previous or concurrent additional malignancy
* Clinically significant pulmonary dysfunction, active infection, prior allogeneic bone marrow transplant, active autoimmune disease
* Positive serology for HIV or hepatitis C
* Hepatitis B surface antigen or hepatitis B core antibody positive
* Pregnant or breastfeeding
* Known current drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | any time point during the study up to 18 months
CLL Cysteine 481 mutation status | CLL patients in Cohort 7 will be followed for 9 months unless no cysteine 481 mutation is detected.
  The primary endpoint for Cohort 7 is the elimination of the cysteine 481 mutant clone (<1%).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | any time point during the study up to 18 months
Progression-free survival (PFS) | any time point during the study up to 18 months
Overall survival (OS) | any time point during the study up to 18 months
Duration of response (DOR) | any time point during the study up to 18 months
Resolution of disease-related symptoms | any time point during the study up to 18 months
  Resolution of disease-related symptoms which are common to the disease include fever, weight loss, night sweats, fatigue, loss of appetite pain, and pruritus; symptoms will be assessed by descriptive statistics and data listings.
Maximum serum drug concentration (Cmax) | any time point during the study up to 12 months
Minimum serum drug concentration (Cmin) | any time point during the study up to 12 months
Area under the concentration-time curve (AUC0-t and AUC0-∞) | any time point during the study up to 12 months
Systemic clearance (CL) | any time point during the study up to 12 months
Volume of distribution (Vd) | any time point during the study up to 12 months
Elimination half-life (t1/2) | any time point during the study up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott C. Stromatt, M.D., Study Director — Aptevo Therapeutics
Locations (8):
- United States (8):
  - Augusta, Georgia
  - Columbus, Ohio
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - Houston, Texas
  - Swedish Cancer Institute,1221 Madison St., Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington